CLINICAL TRIAL: NCT00055835
Title: Phase II Evaluation of Carboplatin, Paclitaxel and Gemcitabine Followed by Concurrent Cisplatin and Radiation Therapy in Patients With Locally Advanced or Recurrent Urothelial Malignancy
Brief Title: S0121, Neoadjuvant Carboplatin, Paclitaxel, and Gemcitabine Followed by Cisplatin and Radiation Therapy in Treating Patients With Locally Advanced or Recurrent Carcinoma of the Urothelium
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: SWOG Cancer Research Network (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000271309; S0121 (Other: SWOG); U10CA032102 (NIH)
Record Dates: First submitted 2003-03-06; First posted 2003-03-07 (Estimated); Last update posted 2013-01-31 (Estimated); Status verified 2013-01

CONDITIONS: Bladder Cancer; Urethral Cancer
Keywords: recurrent bladder cancer; stage III bladder cancer; squamous cell carcinoma of the bladder; stage II bladder cancer; recurrent urethral cancer; urethral cancer associated with invasive bladder cancer; distal urethral cancer; proximal urethral cancer; stage IV bladder cancer; transitional cell carcinoma of the bladder
MeSH Terms: conditions — Urinary Bladder Neoplasms; Urethral Neoplasms | interventions — Carboplatin; Cisplatin; Gemcitabine; Paclitaxel; Neoadjuvant Therapy; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: carboplatin — *AUC=5 (by modified Calvert formula), IV, over 15 minutes; given q 21 days for a maximum of 3 cycles (1 cycle = 21 days)
  Other Names: Paraplatin
Drug: cisplatin — 75 mg/m2 (maximum dose 150 mg), IV, rapid infusion; given q 21 days for 2 cycles (1 cycle = 21 days)
  Other Names: Platinol; CDDP
Drug: gemcitabine hydrochloride — 800 mg/m2, IV, over 30 minutes; given on Days 1 & 8, q 21 days, for a maximum of 3 cycles (1 cycle = 21 days)
  Other Names: Gemzar
Drug: paclitaxel — 200 mg/m2, IV, over 3 hours; given q 21 days for a maximum of 3 cycles (1 cycle = 21 days)
  Other Names: Taxol
Procedure: neoadjuvant therapy — Neoadjuvant chemotherapy (paclitaxel, carboplatin, and gemcitabine)
Radiation: radiation therapy — Radiation treatments will be delivered once daily. Treatment will be given 5 days per week at a dose of 180 to 200 cGy per day. All fields will be treated everyday.

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as carboplatin, paclitaxel, gemcitabine, and cisplatin, work in different ways to stop tumor cells from dividing so they stop growing or die. Radiation therapy uses high-energy x-rays to damage tumor cells. Giving chemotherapy before radiation therapy, and combining chemotherapy with radiation therapy, may kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of neoadjuvant gemcitabine, paclitaxel, and carboplatin followed by cisplatin and radiation therapy in treating patients who have locally advanced or recurrent carcinoma (cancer) of the urothelium.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the overall survival of patients with locally advanced or recurrent carcinoma of the urothelium treated with neoadjuvant carboplatin, paclitaxel, and gemcitabine followed by concurrent cisplatin and radiotherapy.
* Determine the feasibility of administering this regimen to these patients.
* Determine the progression-free survival of patients treated with this regimen.
* Determine the qualitative and quantitative toxic effects of this regimen in these patients.
* Determine the response rate (confirmed and unconfirmed) of patients treated with the neoadjuvant regimen and those treated with the whole regimen.
* Determine the proportion of patients who qualify for concurrent cisplatin and radiotherapy after receiving the neoadjuvant regimen.
* Determine the potential value of suppressor gene expression analysis (p53 and retinoblastoma gene) and HER2 expression as indicators of prognosis and/or response in patients treated with this regimen.

OUTLINE: This is a multicenter study.

Patients receive neoadjuvant chemotherapy comprising paclitaxel IV over 3 hours and carboplatin IV over 15 minutes on day 1 and gemcitabine IV over 30 minutes on days 1 and 8. Treatment repeats every 21 days for a maximum of 3 courses in the absence of disease progression or unacceptable toxicity.

Within 4-8 weeks after the completion of neoadjuvant chemotherapy, patients receive cisplatin IV over 30-60 minutes on day 1. Treatment repeats every 21 days for a maximum of 2 courses in the absence of disease progression or unacceptable toxicity. Patients also undergo concurrent radiotherapy 5 days a week for 6 weeks.

Patients are followed every 3 months for 2 years and then every 6 months for 3 years.

PROJECTED ACCRUAL: A total of 80 patients will be accrued for this study within 4 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed primary or recurrent invasive carcinoma of the urothelium

  * Transitional, squamous, or mixed cell subtypes allowed
  * Primary disease site must be the urinary bladder or urethra
  * Disease confined to the true pelvis (T2-T4, N0-N3, M0)
  * Must meet at least 1 of the following criteria:

    * Nodal involvement at or below the level of the bifurcation of the iliac vessels
    * Medically or surgically inoperable
    * Patient refused cystectomy
* Measurable or nonmeasurable disease
* Evidence of tumor invasion of the muscularis by cystoscopy and biopsy and detailed bladder mapping within the past 56 days
* No extrapelvic metastases
* Eligible to receive radiotherapy

  * Planned radiotherapy at a SWOG-approved facility

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* Zubrod 0-2

Life expectancy

* Not specified

Hematopoietic

* Granulocyte count at least 1,500/mm^3
* Platelet count at least lower limit of normal

Hepatic

* Bilirubin no greater than upper limit of normal (ULN)
* SGOT or SGPT no greater than 2.5 times ULN

Renal

* Creatinine clearance at least 60 mL/min OR
* Creatinine no greater than ULN

Gastrointestinal

* No chronic diarrhea
* No malabsorption
* No extensive diverticular disease of the colon
* No inflammatory bowel disease
* No other pre-existing gastrointestinal disorders

Other

* Not pregnant or nursing
* Fertile patients must use effective contraception
* No active infections requiring antibiotics
* No other malignancy within the past 5 years except adequately treated basal cell or squamous cell skin cancer, carcinoma in situ of the cervix, or adequately treated stage I or II cancer currently in complete remission

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* No prior chemotherapy for patients with a current diagnosis of advanced bladder cancer that is also the initial diagnosis
* No prior systemic chemotherapy except adjuvant therapy for recurrent disease completed more than 6 months ago
* No prior carboplatin
* No prior paclitaxel
* No prior gemcitabine

Endocrine therapy

* Not specified

Radiotherapy

* See Disease Characteristics
* No prior pelvic radiotherapy

Surgery

* See Disease Characteristics
* Recovered from prior surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2002-11; Primary Completion 2006-06 (Actual); Study Completion 2006-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ulka N. Vaishampayan, MD, Study Chair — Barbara Ann Karmanos Cancer Institute
Locations (92):
- United States (92):
  - MBCCOP - Gulf Coast, Mobile, Alabama
  - CCOP - Western Regional, Arizona, Phoenix, Arizona
  - Veterans Affairs Medical Center - Phoenix (Carl T. Hayden), Phoenix, Arizona
  - Veterans Affairs Medical Center - Tucson, Tucson, Arizona
  - Arizona Cancer Center at University of Arizona Health Sciences Center, Tucson, Arizona
  - Arkansas Cancer Research Center at University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Veterans Affairs Medical Center - Little Rock, Little Rock, Arkansas
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - USC/Norris Comprehensive Cancer Center and Hospital, Los Angeles, California
  - Jonsson Comprehensive Cancer Center at UCLA, Los Angeles, California
  - Veterans Affairs Outpatient Clinic - Martinez, Martinez, California
  - CCOP - Bay Area Tumor Institute, Oakland, California
  - Chao Family Comprehensive Cancer Center at University of California Irvine Medical Center, Orange, California
  - University of California Davis Cancer Center, Sacramento, California
  - CCOP - Santa Rosa Memorial Hospital, Santa Rosa, California
  - University of Colorado Cancer Center at University of Colorado Health Sciences Center, Aurora, Colorado
  - Veterans Affairs Medical Center - Denver, Denver, Colorado
  - MBCCOP - Howard University Cancer Center, Washington D.C., District of Columbia
  - Veterans Affairs Medical Center - Tampa (Haley), Tampa, Florida
  - CCOP - Atlanta Regional, Atlanta, Georgia
  - MBCCOP - Hawaii, Honolulu, Hawaii
  - MBCCOP - University of Illinois at Chicago, Chicago, Illinois
  - Veterans Affairs Medical Center - Chicago Westside Hospital, Chicago, Illinois
  - CCOP - Central Illinois, Decatur, Illinois
  - Veterans Affairs Medical Center - Hines, Hines, Illinois
  - Cardinal Bernardin Cancer Center at Loyola University Medical Center, Maywood, Illinois
  - Kansas Masonic Cancer Research Institute at the University of Kansas Medical Center, Kansas City, Kansas
  - CCOP - Wichita, Wichita, Kansas
  - Veterans Affairs Medical Center - Wichita, Wichita, Kansas
  - Veterans Affairs Medical Center - Lexington, Lexington, Kentucky
  - Markey Cancer Center at University of Kentucky Chandler Medical Center, Lexington, Kentucky
  - MBCCOP - LSU Health Sciences Center, New Orleans, Louisiana
  - Tulane Cancer Center at Tulane University Hospital and Clinic, New Orleans, Louisiana
  - Veterans Affairs Medical Center - New Orleans, New Orleans, Louisiana
  - Veterans Affairs Medical Center - Shreveport, Shreveport, Louisiana
  - Feist-Weiller Cancer Center at Louisiana State University Health Sciences, Shreveport, Louisiana
  - Cancer Research Center at Boston Medical Center, Boston, Massachusetts
  - CCOP - Michigan Cancer Research Consortium, Ann Arbor, Michigan
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Veterans Affairs Medical Center - Detroit, Detroit, Michigan
  - Josephine Ford Cancer Center at Henry Ford Health System, Detroit, Michigan
  - CCOP - Grand Rapids, Grand Rapids, Michigan
  - CCOP - Beaumont, Royal Oak, Michigan
  - Providence Cancer Institute at Providence Hospital - Southfield Campus, Southfield, Michigan
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Veterans Affairs Medical Center - Jackson, Jackson, Mississippi
  - CCOP - Kansas City, Kansas City, Missouri
  - CCOP - Cancer Research for the Ozarks, Springfield, Missouri
  - Saint Louis University Cancer Center, St Louis, Missouri
  - CCOP - St. Louis-Cape Girardeau, St Louis, Missouri
  - CCOP - Montana Cancer Consortium, Billings, Montana
  - Veterans Affairs Medical Center - Albuquerque, Albuquerque, New Mexico
  - MBCCOP - University of New Mexico HSC, Albuquerque, New Mexico
  - Western New York Urology Associates, Buffalo, New York
  - NYU Cancer Institute at New York University Medical Center, New York, New York
  - Herbert Irving Comprehensive Cancer Center at Columbia University, New York, New York
  - James P. Wilmot Cancer Center at University of Rochester Medical Center, Rochester, New York
  - CCOP - Southeast Cancer Control Consortium, Goldsboro, North Carolina
  - Veterans Affairs Medical Center - Cincinnati, Cincinnati, Ohio
  - Charles M. Barrett Cancer Center at University Hospital, Cincinnati, Ohio
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - CCOP - Columbus, Columbus, Ohio
  - Veterans Affairs Medical Center - Dayton, Dayton, Ohio
  - CCOP - Dayton, Dayton, Ohio
  - Oklahoma University Medical Center, Oklahoma City, Oklahoma
  - Cancer Institute at Oregon Health and Science University, Portland, Oregon
  - CCOP - Columbia River Oncology Program, Portland, Oregon
  - Veterans Affairs Medical Center - Charleston, Charleston, South Carolina
  - Hollings Cancer Center at Medical University of South Carolina, Charleston, South Carolina
  - CCOP - Greenville, Greenville, South Carolina
  - CCOP - Upstate Carolina, Spartanburg, South Carolina
  - University of Tennessee Cancer Institute at Methodist Central Hospital, Memphis, Tennessee
  - Harrington Cancer Center, Amarillo, Texas
  - Texas Tech University Health Sciences Center School of Medicine, Amarillo, Texas
  - Veterans Affairs Medical Center - Amarillo, Amarillo, Texas
  - Brooke Army Medical Center, Fort Sam Houston, Texas
  - University of Texas Medical Branch, Galveston, Texas
  - M.D. Anderson Cancer Center at University of Texas, Houston, Texas
  - Baylor College of Medicine, Houston, Texas
  - UMC Southwest Cancer and Research Center, Lubbock, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Veterans Affairs Medical Center - San Antonio (Murphy), San Antonio, Texas
  - Veterans Affairs Medical Center - Temple, Temple, Texas
  - CCOP - Scott and White Hospital, Temple, Texas
  - Huntsman Cancer Institute at University of Utah, Salt Lake City, Utah
  - Veterans Affairs Medical Center - Salt Lake City, Salt Lake City, Utah
  - Sentara Cancer Institute at Sentara Norfolk General Hospital, Norfolk, Virginia
  - CCOP - Virginia Mason Research Center, Seattle, Washington
  - Veterans Affairs Medical Center - Seattle, Seattle, Washington
  - Puget Sound Oncology Consortium, Seattle, Washington
  - CCOP - Northwest, Tacoma, Washington